CLINICAL TRIAL: NCT01905891
Title: Nanocytology Evaluation of Epidermal Cells to Assess Risk of Squamous Cell Carcinoma and Field Cancerization in High Risk Patients
Brief Title: Nanocytology Test to Evaluate Skin Cancer in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Joan Guitart, MD, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JG05012013
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Actinic Keratosis; Squamous Cell Carcinoma
Keywords: Non melanoma skin cancer; Field of cancerization; Skin carcinogenesis
MeSH Terms: conditions — Keratosis, Actinic; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects at risk of skin cancer (Other): Subjects at risk of skin cancer (sun-damaged skin) a superficial shave biopsy will be performed.
  Interventions: Procedure: Superficial shave biopsy
- Subjects with healthy skin (Other): Subjects without sun-damaged skin a superficial shave biopsy will be performed.
  Interventions: Procedure: Superficial shave biopsy

INTERVENTIONS:
Procedure: Superficial shave biopsy — Sample will be obtained from random dorsal forearm skin sites without evidence of keratotic lesions. The site will be selected by the investigator. Skin will first be wiped with an alcohol pad and 1% lidocaine will be superficially infiltrated per standard skin surgical procedures. 30% trichloroacetic acid (TCA, standard chemical peel) will then be applied for five minutes. TCA will be neutralized using bicarbonate. Using a cytology brush (a small brush which is used to collect cells during the course of a biopsy) cells will be collected by gentle scraping surface of the skin. Then, a superficial shave biopsy specimen, obtained by using a dermablade (a flexible, one piece blade specifically designed for shave biopsy and excision of skin lesions) will be obtained.

SUMMARY:
The purpose of this study is to correlate pathological features from specimens in order to determine if this new molecular diagnostic technique can be used to detect risk of skin cancer.

DETAILED DESCRIPTION:
Squamous cell carcinoma is the culmination of a multistep carcinogenesis process that is preceded by early stages referred as squamous dysplasia and actinic keratosis. Squamous dysplasia (SD) also known as "field effect" is clinically characterized by xerosis (dry, scaly skin), lentigines and uneven pigmentation. While morphologically skin biopsies and cytology samples show only minimal changes, at the molecular level it is known that SD is characterized by small clone keratinocytes carrying mutations of the P53 gene. An optical technology called Partial Wave Spectroscopy (PWS) probes nanoscale structures in the order of tens to a few hundred nanometers. PWS is a light back-scattering techniques that uses light reflected off of a tissue sample. The measured biomarker is sensitive to the cytosolic and nucleic architecture within the cell and quantifies the nanoscale disorder, which conventional light microscopy fails to appreciate. PWS has allowed to identify various grades of structural disorder at the nanoscale level of colonic and pulmonary premalignant cell samples. Using PWS we aim to study the spectrum of cutaneous SD from patients at high risk for SCC development. Since squamous dysplasia is difficult to assess with routine histology and cytopathology and a grading system for squamous dysplasia by routine histology or cytology is not available, we propose to assess the value of PWS as a new and more sensitive imaging technique. By identifying the degree of SD at the molecular level, we may be able to intervene with close surveillance, early treatment and chemoprevention strategies to achieve lower morbidity by means of fewer and smaller skin cancers.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 89 years old, male and female, Fitzpatrick skin phototype I - III
* Photodamage skin grades 3 - 4 (global assessment)
* Medical history of precancerous lesions and or known history of SCC or healthy volunteers

Exclusion Criteria:

* Subjects under 18 years old
* Pregnant women or lactating mothers
* Treatment with systemic chemotherapy within 4 weeks period before consent
* Known HIV+ patients (self-reported)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Nanocytology assessment of skin cancer risk | 1 year
  The primary outcome measure is to correlate clinical phenotype (age, skin phototype, level of photodamage, history of prior skin cancers) with morphology and nuclear characteristics, in order to determine if this new molecular diagnostic technique can be used to detect early stages of skin carcinogenesis and identify high risk-patients.

SECONDARY OUTCOMES:
Compare nanocytology assessment with pathological findings | 1 year
  Secondary outcome measure is to compare PWS results and clinical phenotype with the evaluation of skin samples by routine cytology/pathology, as they relate to the clinical level of overall photodamaged and prior history of skin cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Guitart, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States